CLINICAL TRIAL: NCT03989102
Title: Randomized, Placebo-Controlled, Double-Blind Study to Assess Safety, Immunogenicity, and Protective Efficacy of Radiation Attenuated Plasmodium Falciparum NF54 Sporozoites (PfSPZ Vaccine) During Malaria Transmission Season in Healthy African Adult Women of Childbearing Potential in Mali
Brief Title: Safety, Immunogenicity, and Protective Efficacy of Radiation Attenuated Plasmodium Falciparum NF54 Sporozoites (PfSPZ Vaccine) During Malaria Transmission Season in Healthy African Adult Women of Childbearing Potential in Mali
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999919113; 19-I-N113
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2022-05

CONDITIONS: Malaria
Keywords: Pregnancy; Tolerability; Immune; Response; Vaccination
MeSH Terms: conditions — Malaria | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Arm 1: (n= 100) will receive 3 doses of PfSPZ Vaccine (9 x10(5)) via direct venous inoculation (DVI) at 1, 8, 29 days.
  Interventions: Biological: PfSPZ Vaccine
- Arm 2 (Experimental): Arm 2: (n= 100) will receive 3 doses of PfSPZ Vaccine (1.8 x10(6)) via DVI at 1, 8, 29 days.
  Interventions: Biological: PfSPZ Vaccine
- Arm 3 (Placebo Comparator): Arm 3: (n=100): will receive 3 doses of normal saline (placebo) injection via DVI at 1, 8, 29 days.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — PfSPZ vaccine is comprised of aseptic, metabolically active, non-replicating, purified, cryopreserved P. falciparum sporozoites.
  Arms: Arm 1; Arm 2
Other: Normal Saline — Sterile isotonic (0.9%) normal saline is a clear liquid, making it indistinguishable from the study product when drawn up into a syringe; and will be used as a placebo, rather than a comparator vaccine
  Arms: Arm 3

SUMMARY:
Background:

Malaria is a disease spread by mosquitos. Pregnant women are highly susceptible to malaria. This can lead to poor health outcomes for pregnant women and their babies. Researchers want to test a malaria vaccine in women of child bearing potential (WOCBP) and pregnant women. This has not been done before.

Objective:

To assess the safety and tolerability of PfSPZ vaccine in healthy Malian WOCBP.

Eligibility:

Healthy women ages 18 38 who live in Ouelessebougou, Mali, and surrounding villages

Design:

Participants will be screened with:

* Physical exam
* Medical history
* Blood, urine, and heart tests
* Multiple-choice test about malaria

Participants will get 3 injections by needle into a vein of the study vaccine or a placebo. All 3 will be within 1 month. They will not know whether they receive the vaccine or placebo.

Participants will receive treatment to prevent malaria. This will be about 2 weeks before the first and third injections.

After the third injection, participants will be followed for about 1 year. They will be tested to see if the vaccine is safe and protects against malaria infection. They will have blood tests.

If participants get a rash or injection site reaction, photos of the site may be taken.

Any women who become pregnant during the trial will be followed through the end of pregnancy. Babies and their mothers will be followed through the first year of life

DETAILED DESCRIPTION:
Pregnant women are highly susceptible to Plasmodium falciparum malaria, leading to substantial maternal, perinatal, and infant mortality. While malaria vaccine development has made significant progress in recent years, no trials of malaria vaccines have ever been conducted in only women of child bearing potential (WOCBP) or in pregnant women.

PfSPZ Vaccine (Sanaria, Inc) is an advanced malaria candidate being developed for use in

pregnant women, owing in part to its highly favorable safety profile. The vaccine is comprised of aseptic, metabolically active, non-replicating, purified, cryopreserved P. falciparum sporozoites. In multiple double-blind, placebo-controlled trials, there have been no differences in adverse events between vaccinees versus controls. PfSPZ Vaccine induces immune responses to the sporozoite and liver stages of parasite development in the human host and prevents progression to blood stage parasitemia as well as averting disease sequelae; a compelling rationale to test PfSPZ Vaccine for its benefits in this proposed population.

Sanaria has already achieved vaccine efficacy against homologous and heterogenous parasite populations in endemic areas following three doses of PfSPZ Vaccine in several studies with 9.0x10^5 and 1.8x10^6 PfSPZ Vaccine and has explored accelerated regimens, such as 1, 8, 29 days. Accelerated PfSPZ Vaccine regimens such as this could induce protection earlier in pregnancy, minimizing the period at risk and improving pregnancy outcomes over the control group.

Given this, the Malaria Research and Training Center, the Laboratory of Malaria Immunology

and Vaccinology National Institute of Allergy and Infectious Diseases, and Sanaria, Inc. propose to initiate testing of the day 1, 8, and 29 dosing regimen of PfSPZ Vaccine in WOCBP, and in subsequent studies, in pregnant women, using doses of 9.0x10^5 and 1.8x10^6 PfSPZ Vaccine. This will be the first step in a clinical development plan for PfSPZ Vaccine in WOCBP and pregnant women: 1) safety and efficacy studies in non-pregnant WOCBP (this trial), 2) studies of the safety and efficacy of a primary immunization series in all trimesters, and 3) studies to evaluate the safety and efficacy of boosting during pregnancy.

A pregnancy registry study (#17-I-N018) has been ongoing in Mali since 2017 to gain

background data on maternal/fetal outcomes in the target population in anticipation of this study. Women who become pregnant during the course of this study, and their offspring, will be followed for maternal clinical outcomes and malaria infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Females of child bearing potential aged greater than or equal to 18 and less than or equal to 38 years
  2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
  3. In good general health and without clinically significant medical history
  4. Willing to have blood samples stored for future research
  5. Available for the duration of the study
  6. Must be willing to use reliable contraception (defined as: pharmacologic contraceptives [parental delivery] or pre-existing intrauterine or implantable device) from 21 days prior to study day 1 to 28 days after last vaccination
  7. Report being interested in becoming pregnant within the next 1-2 years

EXCLUSION CRITERIA:

1. Pregnancy at the time of enrollment/vaccination, as determined by a positive urine or serum human chorionic gonadotropin (beta-hCG) test
2. Biologically unable to become pregnant secondary to: surgical sterilization, premature ovarian insufficiency (defined as no menses for greater than or equal to 12 months without an alternative medical cause)
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
4. Hemoglobin (Hgb), white blood cell count (WBC), absolute neutrophils, and platelets outside the local laboratory-defined limits of normal and greater than or equal to Grade 2 (subjects may be included at the investigators discretion for not clinically significant abnormal values)
5. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal and greater than or equal to Grade 2 (subjects may be included at the investigators discretion for not clinically significant abnormal values)
6. Infected with human immunodeficiency virus (HIV)
7. Known or documented sickle cell disease by history (Note: known sickle cell trait is NOT exclusionary)
8. Clinically significant abnormal electrocardiogram (ECG) such as abnormal corrected QT interval (QTc).
9. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis
10. History of receiving any investigational product within the past 30 days
11. Participation or planned participation in a clinical trial with an investigational product prior to completion of the follow-up visit 28 days following last vaccination OR planned participation in an investigational vaccine study until the last required protocol visit
12. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
13. History of a severe allergic reaction (Grade 2 or higher or per PI discretion) or anaphylaxis
14. Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past two years, or that has required the use of oral or parenteral corticosteroids at any time during the past two years)
15. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren s syndrome, or autoimmune thrombocytopenia
16. Known immunodeficiency syndrome
17. Known asplenia or functional asplenia
18. Use of chronic (greater than or equal to 14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone greater than or equal to 20 mg/day) or immunosuppressive drugs within 30 days of vaccination
19. Receipt of a live vaccine within the past four weeks or a killed vaccine within the past two weeks prior to Vaccination #1 and every subsequent vaccination day
20. Receipt of immunoglobulins and/or blood products within the past six months
21. Previous receipt of an investigational malaria vaccine in the last five years
22. Known allergies or other contraindications against use of artemeter/lumefantrine
23. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol

Max Age: 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 324 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Ouelessebougou Health Research Unit, Wolossébougou, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949
- [Background] Sissoko MS, Healy SA, Katile A, Omaswa F, Zaidi I, Gabriel EE, Kamate B, Samake Y, Guindo MA, Dolo A, Niangaly A, Niare K, Zeguime A, Sissoko K, Diallo H, Thera I, Ding K, Fay MP, O'Connell EM, Nutman TB, Wong-Madden S, Murshedkar T, Ruben AJ, Li M, Abebe Y, Manoj A, Gunasekera A, Chakravarty S, Sim BKL, Billingsley PF, James ER, Walther M, Richie TL, Hoffman SL, Doumbo O, Duffy PE. Safety and efficacy of PfSPZ Vaccine against Plasmodium falciparum via direct venous inoculation in healthy malaria-exposed adults in Mali: a randomised, double-blind phase 1 trial. Lancet Infect Dis. 2017 May;17(5):498-509. doi: 10.1016/S1473-3099(17)30104-4. Epub 2017 Feb 16. PMID 28216244
- [Background] Hoffman SL, Billingsley PF, James E, Richman A, Loyevsky M, Li T, Chakravarty S, Gunasekera A, Chattopadhyay R, Li M, Stafford R, Ahumada A, Epstein JE, Sedegah M, Reyes S, Richie TL, Lyke KE, Edelman R, Laurens MB, Plowe CV, Sim BK. Development of a metabolically active, non-replicating sporozoite vaccine to prevent Plasmodium falciparum malaria. Hum Vaccin. 2010 Jan;6(1):97-106. doi: 10.4161/hv.6.1.10396. Epub 2010 Jan 21. PMID 19946222
- [Background] Sirima SB, Ouedraogo A, Tiono AB, Kabore JM, Bougouma EC, Ouattara MS, Kargougou D, Diarra A, Henry N, Ouedraogo IN, Billingsley PF, Manoj A, Abebe Y, Kc N, Ruben A, Richie TL, James ER, Joshi S, Shrestha B, Strauss K, Lyke KE, Plowe CV, Potter GE, Cox C, Jones W, Sim BKL, Hoffman SL, Laurens MB. A randomized controlled trial showing safety and efficacy of a whole sporozoite vaccine against endemic malaria. Sci Transl Med. 2022 Dec 7;14(674):eabj3776. doi: 10.1126/scitranslmed.abj3776. Epub 2022 Dec 7. PMID 36475905
- [Background] Mordmuller B, Sulyok Z, Sulyok M, Molnar Z, Lalremruata A, Calle CL, Bayon PG, Esen M, Gmeiner M, Held J, Heimann HL, Woldearegai TG, Ibanez J, Flugge J, Fendel R, Kreidenweiss A, Kc N, Murshedkar T, Chakravarty S, Riyahi P, Billingsley PF, Church LWP, Richie TL, Sim BKL, Hoffman SL, Kremsner PG. A PfSPZ vaccine immunization regimen equally protective against homologous and heterologous controlled human malaria infection. NPJ Vaccines. 2022 Aug 23;7(1):100. doi: 10.1038/s41541-022-00510-z. PMID 35999221
- [Background] Sissoko MS, Healy SA, Katile A, Zaidi I, Hu Z, Kamate B, Samake Y, Sissoko K, Mwakingwe-Omari A, Lane J, Imeru A, Mohan R, Thera I, Guindo CO, Dolo A, Niare K, Koita F, Niangaly A, Rausch KM, Zeguime A, Guindo MA, Bah A, Abebe Y, James ER, Manoj A, Murshedkar T, Kc N, Sim BKL, Billingsley PF, Richie TL, Hoffman SL, Doumbo O, Duffy PE. Safety and efficacy of a three-dose regimen of Plasmodium falciparum sporozoite vaccine in adults during an intense malaria transmission season in Mali: a randomised, controlled phase 1 trial. Lancet Infect Dis. 2022 Mar;22(3):377-389. doi: 10.1016/S1473-3099(21)00332-7. Epub 2021 Nov 18. PMID 34801112
- [Derived] Diawara H, Healy SA, Mwakingwe-Omari A, Issiaka D, Diallo A, Traore S, Soumbounou IH, Gaoussou S, Zaidi I, Mahamar A, Attaher O, Fried M, Wylie BJ, Mohan R, Doan V, Doritchamou JYA, Dolo A, Morrison RD, Wang J, Hu Z, Rausch KM, Zeguime A, Murshedkar T, Kc N, Sim BKL, Billingsley PF, Richie TL, Hoffman SL, Dicko A, Duffy PE; PfSPZ Vaccine Study Team. Safety and efficacy of PfSPZ Vaccine against malaria in healthy adults and women anticipating pregnancy in Mali: two randomised, double-blind, placebo-controlled, phase 1 and 2 trials. Lancet Infect Dis. 2024 Dec;24(12):1366-1382. doi: 10.1016/S1473-3099(24)00360-8. Epub 2024 Aug 14. PMID 39153490

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 324 participants were enrolled, but 24 participants were not assigned to any treatment arms due to withdrawn consent; thus 300 total participants were assigned to treatment arms.
Groups:
- Arm 1: 9x10^5 Dose: Participants received 3 doses of PfSPZ Vaccine (9 x10^5) via direct venous inoculation (DVI) at 1, 8, 29 days. Oral antimalarial treatment with artemether/lumefantrine (AL) was given 2 weeks prior to 1st and 3rd injection.
- Arm 2: 1.8 x 10^6 Dose: Participants received 3 doses of PfSPZ Vaccine (1.8 x10^6) via direct venous inoculation (DVI) at 1, 8, 29 days. Oral antimalarial treatment with artemether/lumefantrine (AL) was given 2 weeks prior to 1st and 3rd injection.
- Arm 3: Placebo Comparator: Participants received 3 doses of saline injection via direct venous inoculation (DVI) at 1, 8, 29 days. Oral antimalarial treatment with artemether/lumefantrine (AL) was given 2 weeks prior to 1st and 3rd injection.
Period: Year 1
Arm/Group | Arm 1: 9x10^5 Dose | Arm 2: 1.8 x 10^6 Dose | Arm 3: Placebo Comparator
Started | 100 | 100 | 100
Completed | 88 | 96 | 87
Not Completed | 12 | 4 | 13
Not completed — Withdrawal by Subject | 6 | 2 | 7
Not completed — Lost to Follow-up | 5 | 2 | 5
Not completed — Subject met withdrawal criteria | 1 | 0 | 1
Period: Year 2
Arm/Group | Arm 1: 9x10^5 Dose | Arm 2: 1.8 x 10^6 Dose | Arm 3: Placebo Comparator
Started | 85 | 92 | 84
Completed | 66 | 78 | 68
Not Completed | 19 | 14 | 16
Not completed — Lost to Follow-up | 7 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Subject non-compliant | 3 | 2 | 0
Not completed — Travel | 1 | 0 | 1
Not completed — P16 missing | 4 | 2 | 1
Not completed — P11 missing | 1 | 3 | 7
Not completed — Definitive displacement outside the study site | 0 | 1 | 0
Not completed — Subject missed last study visit | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Subject not reachable | 0 | 0 | 1
Period: Post-Year 3 (up to 3 Years, 8 Months)
Arm/Group | Arm 1: 9x10^5 Dose | Arm 2: 1.8 x 10^6 Dose | Arm 3: Placebo Comparator
Started | 68 | 79 | 71
Completed | 63 | 72 | 67
Not Completed | 5 | 7 | 4
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Widowhood | 1 | 0 | 0
Not completed — Missed last study visit | 2 | 1 | 0
Not completed — Travel | 0 | 3 | 0
Not completed — Relocated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Participants received 3 doses of PfSPZ Vaccine (9 x10^5) via direct venous inoculation (DVI) at 1, 8, 29 days. Oral antimalarial treatment with artemether/lumefantrine (AL) was given 2 weeks prior to 1st and 3rd injection.
- Arm 2: Participants received 3 doses of PfSPZ Vaccine (1.8 x10^6) via direct venous inoculation (DVI) at 1, 8, 29 days. Oral antimalarial treatment with artemether/lumefantrine (AL) was given 2 weeks prior to 1st and 3rd injection.
- Arm 3: Participants received 3 doses of saline injection via direct venous inoculation (DVI) at 1, 8, 29 days. Oral antimalarial treatment with artemether/lumefantrine (AL) was given 2 weeks prior to 1st and 3rd injection.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 100 | 300
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 100 | 300
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Bambara | 72 | 76 | 74 | 222
  Dogon | 1 | 0 | 0 | 1
  Kakolo | 2 | 1 | 0 | 3
  Koroko | 1 | 0 | 0 | 1
  Malinke | 4 | 4 | 3 | 11
  Peulh | 7 | 7 | 10 | 24
  Sarakole | 8 | 5 | 4 | 17
  Senoufo | 1 | 1 | 0 | 2
  Soninke | 3 | 1 | 6 | 10
  Sonrhai | 1 | 1 | 0 | 2
  Bobo | 0 | 1 | 1 | 2
  Gana | 0 | 1 | 0 | 1
  Mossi | 0 | 1 | 1 | 2
  Wolof | 0 | 1 | 0 | 1
  Mianka | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Mali | 100 | 100 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Within 7 Days After Each Vaccine Administration
Description: Assess safety and tolerability of PfSPZ Vaccine primary series in healthy Malian women of child-bearing potential (WOCBP) when given at 1, 8, 29 days at two doses (9 x10^5; 1.8 x10^6).
Time Frame: 7 days after each vaccination at days 1, 8, and 29
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 100 | 100 | 100
Participants | 51 | 43 | 43

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed for 7 days after each vaccination at days 1, 8, and 29, All-Cause Mortality monitored/assessed through year 4
Arm/Group | Arm 1 | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 51/100 | 43/100 | 43/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=100) | Arm 2 (N=100) | Arm 3 (N=100)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 28 (35) | 25 (27) | 26 (31)
Hemoglobin decreased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 2 (2) | 2 (2)
Injection site edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 7 (9) | 6 (6) | 8 (9)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Neutrophil count decreased (Investigations) | 4 (5) | 5 (5) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pruritus (localized) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritis (generalized) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 4 (4) | 5 (6) | 3 (3)
White blood cell count increased (Investigations) | 0 (0) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT03989102/Prot_SAP_000.pdf